CLINICAL TRIAL: NCT04065126
Title: Physical Activity Intervention for Trauma Afflicted Refugees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Red Cross University College (Other)
Collaborators: Swedish Red Cross (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/1174-31
Record Dates: First submitted 2019-05-02; First posted 2019-08-22 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: PTSD; Depression, Anxiety; Physical Activity
Keywords: Mental health; Physical activity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Motor Activity; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity Intervention (Experimental): This arm receives ten two-hour group sessions with physical activity and psycho-educational components, held by a physiotherapist over a period of ten weeks.
  Interventions: Behavioral: Physical activity intervention
- Brief Psycho-education (Active Comparator): This arm receives two brief lectures of psycho-education held by a physiotherapist.
  Interventions: Behavioral: Brief psycho-education

INTERVENTIONS:
Behavioral: Physical activity intervention — Ten sessions (two hours each) with physical activity and psycho-educational components.
  Arms: Physical activity Intervention
Behavioral: Brief psycho-education — Two brief lectures with psycho-educational components, soon after baseline assessment and in connection to follow-up assessment.
  Arms: Brief Psycho-education

SUMMARY:
This study evaluates the effects of a 10-session physical activity intervention for trauma afflicted refugees. Half of participants will receive this 10-session physical activity intervention and half of the participants will be allocated to the control group.

DETAILED DESCRIPTION:
Physical activity, particularly when performed in social settings, has been found to constitute an effective stress reliever and has been associated with improved physical and mental well-being, functional capacity and overall life satisfaction, as well as decreased risk of lifestyle diseases in various populations. Physical activity can also revert symptoms of psychiatric disorders such as depression, anxiety, social isolation and dissociation, which is common among trauma afflicted refugees. Many refugees also suffer from PTSD, and so the investigator's aim is to evaluate what effect a 10-session physical activity intervention will have on the mental and physical health of trauma afflicted refugees in a northern European country. The sessions will include physical exercise as well as psychoeducational components, and will be held by a physiotherapist over a period of ten weeks. The physical activity intervention group will be compared to a control-group, who receives two brief lectures on psycho-education in connection to baseline-assessment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Arabic/Persian speaking persons.
* Persons with refugee background referred to the Swedish Red Cross Treatment Center for trauma related to war and/or torture.
* Person able to undertake physical activity in a group setting.

Exclusion Criteria:

* Current serious suicidal ideation, psychosis, serious cognitive impairments, current substance abuse, acute physical injuries or other health conditions that constrain physical activity.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in symptoms of PTSD | Baseline, 10 weeks, and six months
  Change in symptoms of PTSD measured by the Posttraumatic Stress Disorder Checklist for DSM-V (PCL-5). The PCL-5 is a self-report questionnaire comprising 20 items relating to the main symptoms of PTSD, and which may be divided into the four symptom clusters of PTSD; intrusion, hyperarousal/reactivity, avoidance, and negative alterations in cognitions and mood. Scores range between 0-80. Higher score indicate worse outcome. Initial research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD across samples.

SECONDARY OUTCOMES:
Emotional distress | Baseline, 10 weeks, and six months
  Change in emotional distress (depression and anxiety) assessed by the Hopkins Symptom Checklist (HSCL-25, 25 items). HSCL-25 consists of 10 anxiety and 15 depression items. The items, which refer to how specific symptoms have bothered or distressed the individual during the last week, have four response alternatives ranging from 'not at all' (1) to 'very much' (4). Individual mean item scores will be calculated separately for the anxiety and depression subscales. Respondents with a mean item score above 1.80 and 1.75 classifies as having depression or anxiety, respectively.
Subjective well-being | Baseline, 10 weeks, and six months
  Change in subjective well-being (SWB) assessed by WHO-5 Well-being Index (WHO-5) (5 items). WHO-5 contains five statements of the type 'I have felt happy and in a good mood' and the response alternatives range from 'all the time' (5) to 'never' (0) in relation to the last 2 weeks. The highest possible value of that scale is 100, as the total score is multiplied by a factor of four. Those with values below 50 are classified as having low SWB.
Health related quality of life | Baseline, 10 weeks, and six months
  Change in general health, health-related quality of life, assessed by the EuroQol 5 dimenstions, 5 levels (EQ-5D-5L) (5 items). This instrument consists of a descriptive system including the following five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The respondent's answer on each of the five dimensions results in a one-digit number indicating the level selected for that dimension. The digits for the five dimensions are combined in a five-digit number describing the respondent's health state. The health states may be converted into a single index value between zero and one, where zero being equal to death and one being equal to a state of perfect health.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Saboonchi, Professor, Principal Investigator — Swedish Red Cross University College
Locations (1):
- The Swedish Red Cross Treatment Center for Persons affected by War and Torture (SRCTC), Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No